CLINICAL TRIAL: NCT01219751
Title: Phase II Trial Of Sunitinib In Advanced Non-Clear Cell Type Renal Cell Carcinoma
Brief Title: Trial Of Sunitinib In Advanced Non-Clear Cell Type Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Seoul National University Hospital (Other); Kyungpook National University Hospital (Other)
Responsible Party: Jae Lyun Lee/Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UOSG_AMC_0801
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2010-09

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib 50 mg D1-D28 every 6 weeks
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 50 mg D1-D28 every 6 weeks
  Other Names: Sutene

SUMMARY:
To evaluate the efficacy and safety of sunitinib in non-clear cell type renal cell carcinoma with the exception of pure sarcomatoid carcinoma and collecting duct carcinoma

DETAILED DESCRIPTION:
There have been no standard treatment in non-clear cell renal cell carcinoma. Retrospective studies showed sunitinib or sorafenib might be active in non-clear cell renal cell carcinoma, especially papillary type and chromophobe type.

This study is to evaluate efficacy and safety of sunitinib in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmation of renal cell carcinoma without a clear cell histologic component, e.g., papillary type, chromophobe type, or collecting duct type
2. Patients with stage IV or recurrent disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent.
3. Measurable disease according to RECIST criteria
4. ECOG performance status 1 or better
5. Age 18 years or older
6. Adequate cardiac function
7. Adequate bone marrow, hepatic, and renal function
8. Life expectancy of ≥ 3 months
9. Singed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

1. Clear cell type renal cell carcinoma or sarcomatoid carcinoma without any clue to the primary type
2. Diagnosis of any serious secondary malignancy within the last 2 years, except for adequately treated basal cell or squamous cell carcinoma of skin, or in situ carcinoma of cervix uteri
3. Hypertension that cannot be controlled by medications (blood pressure > 150/90 mmHg despite optimal medical therapy)
4. Treatment with anticonvulsant agents and treatment with therapeutic doses of coumadin currently or within 2 weeks prior to first day of sunitinib administration. Low dose coumadin for DVT prophylaxis is permitted (up to 2 mg/day).
5. Pregnancy or breast feeding.
6. Other severe acute or chronic medical or psychiatric condition
7. Prior treatment on sunitinib, sorafenib, or bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Response rate | up to 12 months
  Tumor response is to be measured every 6 weeks. RECIST v.1.1 will be used to definte target lesion and non-target lesion and classify the response category.

SECONDARY OUTCOMES:
Progression free survival | up to 24 months
  Form the date of enrollment to the date of the first documented disease progression or death from any cause, which came first.
overall survival | up to 36 months
Safety | up to 24 months
  Safety will be assessed using CTCAE v.3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Lyun Lee, MD, PhD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee JL, Ahn JH, Lim HY, Park SH, Lee SH, Kim TM, Lee DH, Cho YM, Song C, Hong JH, Kim CS, Ahn H. Multicenter phase II study of sunitinib in patients with non-clear cell renal cell carcinoma. Ann Oncol. 2012 Aug;23(8):2108-2114. doi: 10.1093/annonc/mdr586. Epub 2012 Jan 6. PMID 22228449